CLINICAL TRIAL: NCT07294560
Title: Evaluation of the Effect of Perioperative Recruitment Maneuver Practice on Lung Ultrasound Score and Mechanical Power in Pediatric Patients; A Prospective Randomized Study
Brief Title: Evaluation of the Effect of Perioperative Recruitment Maneuver Practice on Lung Ultrasound Score and Mechanical Power in Pediatric Patients
Acronym: LUS RM PEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Keskin, Elif Keskin, Medical Doctor, Istanbul University - Cerrahpasa, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1408545
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pulmonary Complications; Postoperative Pulmonary Atelectasis; Pediatric Surgery
Keywords: recruitment maneuver; pediatric recruitment maneuver; PEEP; mechanical power; mechanical work; compliance; atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1 (No Intervention): Fixed PEEP: 5 cm H2O
- GROUP 2 (Active Comparator): PEEP: 5 cm H2O, 5 cycles, recruitment maneuver will be performed with pre-extubation plateau P < 35 cm H2O and vital capacity x 2
  Interventions: Other: recruitment maneuver
- GROUP 3 (Active Comparator): PEEP: 5 cm H2O, 5 cycles of recruitment maneuvers will be performed in the right-left lateral decubitus position before extubation with plateauP < 35 cm H2O and vital capacity x 2.
  Interventions: Other: right and left lateral decubitus position recruitment maneuvers

INTERVENTIONS:
Other: recruitment maneuver — PEEP: 5 cmH2O, 5 cycles, recruitment maneuver with plateau P<35 cm H2O and vital capacity x2.
  Arms: GROUP 2
Other: right and left lateral decubitus position recruitment maneuvers — PEEP: 5 cmH2O, 5 cycles of recruitment maneuvers will be performed in the right and left lateral decubitus position before extubation with P<35 cmH2O and vital capacity x2.
  Arms: GROUP 3

SUMMARY:
Pulmonary atelectasis is common during general anesthesia and increases the risk of hypoxemia, especially in pediatric patients. PEEP and recruitment maneuvers (RM) are effective in preventing atelectasis. Lung ultrasound is practical for diagnosis. Mechanical power refers to the amount of energy delivered to the lung by the ventilator; excessive mechanical power can cause lung injury. Limiting mechanical power may reduce postoperative complications. This study aimed to determine the effectiveness of recruitment maneuvers in preventing atelectasis using lung ultrasound during the intraoperative period, to examine the relationship between lung ultrasound scores and mechanical power, and to demonstrate the effect of recruitment maneuvers on postoperative pulmonary complications. This study is based on the hypothesis that "The recruitment maneuver reduces perioperative atelectasis and the development of related complications, and lung ultrasound can be used to detect this. The lung ultrasound score also decreases in patients with reduced mechanical force." It will be prospectively applied to pediatric patients aged 1-14 years who will undergo surgery in the operating rooms of Cerrahpaşa Medical Faculty.

Patients included in the study will be prospectively randomized into 3 groups. The randomization performed using the sealed opaque envelope method.All patients will be ventilated in VG-Pressure guaranteed mode. Tidal volume will be calculated as 6-8 ml/kg of ideal body weight.

GROUP 1: Fixed PEEP: 5 cmH2O, GROUP 2: PEEP: 5 cmH2O, 5 cycles, recruitment maneuver with plateau P<35 cm H2O and vital capacity x2. GROUP 3: PEEP: 5 cmH2O, 5 cycles of recruitment maneuvers will be performed in the right and left lateral decubitus position before extubation with P<35 cmH2O and vital capacity x2.

Lung ultrasound will be performed before induction (1), 5 minutes after intubation (2), before extubation (3), and finally 5 minutes after extubation(4). Each hemithorax will be divided into 6 regions, and lung scores will be recorded. At 5 minutes after intubation and every hour there after, PeakP, PlateauP, DeltaP, Compliance, Driving Pressures, and Mechanical Work calculations will be recorded before and after the maneuver in the group undergoing the recruitment maneuver.

DETAILED DESCRIPTION:
Pulmonary atelectasis refers to incomplete expansion of the alveoli and terminal bronchioles. Atelectasis impairs oxygenation of the blood and reduces lung compliance. Pulmonary atelectasis is common in patients undergoing general anesthesia. The pediatric patientgroup is more sensitive to hypoxemia due to lower functional residual capacity and increased metabolic requirements compared to adults. Therefore, preventing and detecting atelectasis is important. Recruitment maneuvers open collapsed alveoli, increase gas exchange, and improve oxygenation. Lung ultrasound is a fast, simple, non-invasive, and radiation-free technique for diagnosing anesthesia-induced atelectasis. Mechanical work is a recently defined ventilation parameter. This concept represents the energy transferred by the ventilator to the respiratory system per unit time. Part of this energy may directly affect lung tissue, causing ventilator-induced lung injury. Mechanical work is calculated based on a combination of parameters such as tidal volume, respiratory rate, driver pressure, and peak pressure. Mechanical work is a comprehensive measure that reflects the static and dynamic components of these variables together. In intensive care patients, both driving pressure and mechanical power have been shown to be associated with morbidity and mortality. However, in the pediatric patient group, the effect of mechanical power during the intraoperative period on postoperative pulmonary complications has not been sufficiently investigated. Limiting intraoperative mechanical power may reduce the risk of postoperative complications.This study aimed to determine the effectiveness of the recruitment maneuver in preventing atelectasis using lung ultrasound during the intraoperative period, to examine the relationship between the lung ultrasound score and mechanical power, and to demonstrate the effect of the recruitment maneuver on postoperative pulmonary complications.

During the study period, patients aged 1-14 years who underwent surgery in the operating rooms of Cerrahpaşa Medical Faculty, with an ASA score of 1-3, and a surgical duration of at least 2 hours will be included in the study. Patients with an ASA score of 4 or defined lung disease (patients using medication due to asthma and having made 2 emergency visits within 1 year), prematurity (< 36 weeks gestation/bronchopulmonary dysplasia), cystic fibrosis, diagnosed syndromic disease, congenital cardiac disease, abnormal chest X-ray, chest wall deformity, or history of previous chest surgery will be excluded from the study. All patients will be ventilated in VG-Pressure guaranteed mode, Tidal volume will be calculated as ideal body weight x 6-8 ml/kg GROUP 1: Fixed PEEP: 5 cm H2O, GROUP 2: PEEP: 5 cm H2O, 5 cycles, recruitment maneuver will be performed with pre-extubation plateau P < 35 cm H2O and vital capacity x 2

. GROUP 3: PEEP: 5 cm H2O, 5 cycles of recruitment maneuvers will be performed in the right-left lateral decubitus position before extubation with plateauP < 35 cm H2O and vital capacity x 2.

This study will be performed pre-induction (1), 5 minutes after intubation (2), pre-extubation (3), and finally 5 minutes after extubation (4). In the lung ultrasonographic examinations performed, each hemithorax will be divided into 6 regions, and pleural shift, A-line, Air Bronchogram, B score, and Consolidation score will be evaluated at each of the two Plaps points in terms of B score and consolidation score.

Lung scores will be calculated and recorded. Starting from the pre-induction period, at 5 minutes post-intubation and every hour thereafter, KAH, OAB, SpO2, FiO2, ETCO2, Peak P, Plateau P, Delta P, Compliance, driving pressures, mechanical power calculations, and values will be recorded.

Additionally, in groups where the recruitment maneuver is performed, pre- and post-maneuver values will be recorded. Additionally, in groups undergoing recruitment maneuvers, pre- and post-maneuver values will be recorded.

Mechanical power; MPvcv = RR x TV x (PIP - [(Pplat - PEEP) x 0.5]) x 0.098 Dynamic power : (TV x RR x [(Pplato + tPEEP) x 0.5) x 0.098 Driving force: (TV x RR x [ (Pplato - tPEEP) x 0.5] x 0.098 Mechanical Energy (0.098 (TV kg) (PIP -[(Pplato - PEEP) x 0.5] All patients will be premedicated with midazolam (0.05 -1 mg/kg) if vascular access is available, then taken to the operating room. After patients are taken to the operating room, standard monitoring will be performed (SPO2, ECG, and non-invasive blood pressure measurement). Following preoxygenation with 100% O2, induction will be performed with thiopental 5 mg/kg, propofol 2 mg/kg, fentanyl 2 mcg/kg, rocuronium 0.6 mg/kg. After tracheal intubation, the mechanical ventilator will be set to pressure-controlled mode with tidal volume: 8 ml/kg, PEEP: 5 cmH2O, FIO2: 40%, respiratory rate ETCO2: 35-45. Anesthesia maintenance will be provided with sevoflurane/oxygen. 2 mg/kg sugammadex will be used when waking patients. The Aldrete scoring system will be used for service transfer in the recovery unit.

Patients will be monitored for desaturation, fever, and oxygen needs during the 24-hour postoperative period, and findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-14 years with
* ASA score of 1-3
* who had surgery in the operating rooms of Cerrahpaşa Medical Faculty during the study period
* surgical duration was at least 2 hours

Exclusion Criteria:

* ASA score of 4
* defined lung disease (patients using medication due to asthma and having 2 emergency visits within 1 year)
* prematurity (< 36 weeks gestational age / bronchopulmonary dysplasia)
* cystic fibrosis
* diagnosed syndromic disease
* congenital cardiac disease
* abnormal chest X-ray
* chest wall deformity
* or history of previous chest surgery

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Lung Ultrasound Score | perioperative
  The lung ultrasound score will be calculated and recorded before induction, 5 minutes after intubation, before extubation, and 5 minutes after extubation. Lung ventilation loss can be assessed with the LUS Score. This assessment is performed on a total of 12 surfaces, divided by the anterior and posterior axillary lines on the thoracic wall, in the upper and lower parts of the anterior, lateral, and posterior regions. In this scoring system, a score between 0 and 3 is assigned to each of these surfaces. The total score ranges from 0 to 36, and higher scores indicate more severe ventilation loss.
Mechanical Power | perioperative
  Mechanical power calculated using airway pressure, tidal volume, respiratory rate and PEEP parameters to quantify ventilator-induced mechanical energy delivered to the lungs. Mechanical power = RR x TV x (PIP - [(Pplat - PEEP) x 0.5]) x 0.098

SECONDARY OUTCOMES:
postoperative pulmonary complication | postoperative 24 hours
  The secondary outcome is to compare the incidence of clinically significant postoperative pulmonary complications (atelectasis, decreased oxygen saturation, and need for postoperative respiratory support) between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Keskin, Medical Doctor, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No